CLINICAL TRIAL: NCT01402024
Title: A Study to Evaluate the Anti-emetic Effect of Aprepitant Versus Placebo as an Add-on Therapy in Children and Adolescent Receiving Chemotherapy: A Randomized, Doubly Blinded Controlled Trial
Brief Title: Study to Evaluate Anti-emetic Effect of Aprepitant Versus Placebo in Children and Adolescent Receiving Chemotherapy
Acronym: Aprepitant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Principal Investigator, Sameer Bakhshi, Additional Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CT/38/011/RS
Record Dates: First submitted 2011-07-19; First posted 2011-07-26 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant (Experimental): It is an double blind randomized placebo controlled trial with age group of 5-18 years and weight between 15-65 kg, who will receive highly emetogenic chemotherapy. Patient who will meet the inclusion criteria will be randomly enrolled in either of the two arm-aprepitant arm and control arm. The patient on aprepitant arm will receive the study drug (aprepitant)along with standard anti-emetic therapy (as per the dosages mentioned in the protocol).
  Interventions: Drug: Aprepitant
- Control (Placebo Comparator): It is an double blind randomized placebo controlled trial with age group of 5-18 years and weight between 15-65 kg, who will receive highly emetogenic chemotherapy. Patient who will meet the inclusion criteria will be randomly enrolled in either of the two arm-aprepitant arm and control arm. The patient on the control arm will receive the placebo along with standard anti-emetic therapy (as per the dosages mentioned in the protocol).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant — The patient on study group with weight category of 15-40 kg will receive:
  D1- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant 80 mg; D2- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant 80 mg; D3- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant 80 mg and
  The patient with weight category of 41-65 kg in study group will receive:
  D1- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant 125 mg; D2- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant 80 mg; D3- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant 80 mg
  Other Names: Empov
  Arms: Aprepitant
Drug: Placebo — Patient on control group with weight category of 15-40 kg will receive:
  D1- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant placebo 80 mg; D2- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant placebo 80 mg; D3- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant placebo 80 mg; and
  The patient on control group with weight category of 41-65 kg will receive:
  D1- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant placebo 125 mg; D2- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant placebo 80 mg; D3- Dexamethasone 0.15 mg/kg, ondansetron (0.15 mg/kg, single dose), Aprepitant placebo 80 mg (all are injectable except Aprepitant oral capsule).
  Other Names: Empov placebo capsules
  Arms: Control

SUMMARY:
Chemotherapy induced nausea and vomiting (CINV) is one of the few mostly observed distressing toxicity of cancer treatment. It can occur up to 90% in case of highly emetogenic chemotherapy use. CINV causes disturbance in daily living of cancer patient and reduces compliance with treatment Even with the standard anti-emetic measures up to 50% patient can suffer from this complication. Whereas there is standard anti-emetic guideline exists in case of adult patients, there no such guidelines made in pediatric population. The new drug Aprepitant has been recommended for use in adults with high efficacy, there no such concrete data available in children regarding its use. There are few retrospective reports and limited data available regarding use of Aprepitant in children with satisfactory efficacy in reducing CINV. As there no randomized large data to suggests its efficacy and its routine use in children, we have planned this study.

DETAILED DESCRIPTION:
Population:

Children and adolescents (5-18 years) with weight between 15-65 kg receiving highly emetogenic chemotherapy (HEC) -

* VAC (vincristine, dactinomycin/Adriamycin, cyclophosphamide)
* ABVD (adriamycin, bleomycin, vinblastine, dacarbazine)
* Cisplatin/Doxorubicin

Sampling technique Subjects who met the eligibility criteria will be randomly assigned using random allocation number generated by computer into one of the two groups. The unit of randomization will be the subject at first cycle of HEC. The same patient will not be enrolled for twice

Procedure for data collection:

1. The data will be collected from each patient from d1 to d10 of chemotherapy of which patient will received chemotherapy in day care, maximum up to d3.
2. After taking consent patient will be enrolled as per inclusion and exclusion criteria, and randomized to one of two groups. All baseline assessment will be done. Patient will be explained about the filling of the diary. In first 2 days. The subjects will fill the diary under the investigator supervision, and the rest of filling will be in home. Reinforcement will be done over phone.

Procedure of double blinding

* Double blinding will be done for the intervention. Four different boxes will be made for capsules. Total 3 capsules for 3 days will be made in a blister pack, mentioning the d1, d2, d3 (for each capsule). Two different body weight groups will be made: 15-40 kg, and 41-65 kg.
* Group "A" will be the code for Aprepitant group and group "B" will be code for control group. Both patient and the investigator will be blinded regarding medicine in the code.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have a confirmed diagnosis of malignancy and receiving highly emetogenic chemotherapy first time (VAC, ABVD and CDDP/Doxorubicin)
* Age group 5-18 years with weight between 15-65 kg
* Children/adolescents and their caregiver who can understand Hindi or English and willing to participate in the study (with written informed consent)

Exclusion Criteria:

* Significant organ dysfunction
* Active infection
* Pregnancy
* Uncontrolled medical condition other than malignancy
* Need for contraindicated concomitant medication
* Patients receiving chemotherapy other than VAC, ABVD and CDDP/Doxorubicin
* Treatment with another investigational drug within 4 weeks of study start or prior Aprepitant use
* Had received or will receive RT to abdomen or pelvis in the week prior to treatment
* Vomited in the 24 hr prior to treatment
* Prior exposure to highly emetogenic chemotherapeutics
* Abnormal lab values (ANC<1500/mm3, TLC<3000/mm3, Plt<100,000/mm3, AST/ALT> 2.5 times of ULN, bill>1.5 times of ULN, S.cr>1.5 times of ULN, patient on systemic steroids

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
- Numbers of episodes of nausea and vomiting. - Duration of nausea (in hours). - Severity of nausea as per Edmonton's Symptom Assessment System (ESAS), numerical scale for nausea. | 5 days

SECONDARY OUTCOMES:
- Chemotherapy induced additional side effects. - Number of anti-emetic dosage (other than aprepitant) required for treatment of vomiting. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Bakhshi, MD, Principal Investigator — Dr. BRA IRCH, AIIMS, New Delhi (India)
Locations (1):
- Dr. BRA IRCH, AIIMS, New Delhi, National Capital Territory of Delhi, India